CLINICAL TRIAL: NCT06897384
Title: High-dose Intravenous Vitamin C for the Treatment of Severe Acute Pancreatitis
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Shanghai Municipal Science and Technology Commission (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024430
Record Dates: First submitted 2025-02-26; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-10

CONDITIONS: Severe Acute Pancreatitis
Keywords: high-dose intravenous vitamin C; severe acute pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Sodium Chloride; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vitamin C Group (Experimental): The intervention is the administration of vitamin C via central venous infusion at a rate of 500mg/kg/24h, 2g/h, for a total of 7 days.
  Interventions: Drug: Vitamin C (Ascorbic Acid)
- Control Group (Placebo Comparator): The intervention for the control group involves administering the same dosage of normal saline via the same injection method for a total of 7 days.
  Interventions: Drug: Saline (NaCl 0,9 %)

INTERVENTIONS:
Drug: Saline (NaCl 0,9 %) — The control group involves only adding 50ml of normal saline to a 50ml syringe, without any labels to ensure identical appearance, and the method of administration and dosage are the same with vitamin C group.
  Arms: Control Group
Drug: Vitamin C (Ascorbic Acid) — Vitamin C at dose of 500mg/kg/24h, 2g/h
  Other Names: Vitamin C group
  Arms: Vitamin C Group

SUMMARY:
This study is a prospective, randomized, double-blinded, parallel-controlled, multi-central clinical trial for patients with severe acute pancreatitis (SAP). Patients with SAP in the early stage (within 7 days of onset) and over the age of 18, based on the routine treatment, will be randomly divided into a high-dose intravenous vitamin C group (HDIVC, 500mg/kg/24h, administered by iv. pump at a rate of 2g/h for 7 days) and a control group (an equal volume of normal saline). The primary endpoint is mortality rate in ICU, and secondary endpoints include free organ support duration (FOSD) within 14 days after enrollment, changes in inflammatory response and severity, disease severity scores and changes, fluid retention, incidence of infectious pancreatic necrosis (IPN), ICU mortality, pancreatic necrosis scores, monitoring of vitamin C plasma concentrations before and after HDIVC use, composition of gut microbiota, observation of vitamin C-related adverse reactions. The study hypothesis is that HDIVC can reduce mortality rate in ICU, significantly decrease the FOSD within 14 days and significantly reduce inflammatory response, decrease fluid retention, and improve disease severity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Time from onset of illness to enrollment is less than 7 days
* Meet the 2012 Atlanta Guidelines SAP diagnostic criteria

Exclusion Criteria:

* SAP caused by tumors or ERCP
* Pregnant or breastfeeding
* Allergic to vitamin C
* Use of other experimental drugs within the timeframe of this study
* Chronic organs failure such as heart, liver, lung, or kidney before admission, with specific indicators being (chronic cardiovascular dysfunction requiring long-term mechanical hemodynamic support or inotropic drug support; chronic obstructive pulmonary disease requiring home oxygen therapy; chronic liver dysfunction at Child-Pugh Class C; chronic kidney disease with an estimated glomerular filtration rate (eGFR) of less than 60 mL/min/1.73 m² or serum creatinine greater than 150 μmol/L)
* Immunosuppressed state, including malignant tumors, post-transplant status, long-term use of immunosuppressor (for at least 1 month before enrollment), AIDS, etc.
* The patient and family are unwilling to sign the informed consent form
* Body weight greater than 100kg
* Urinary system stones

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality rate in ICU | through study completion, an average of 6 months

SECONDARY OUTCOMES:
The Impact of HDIVC on Free Organ Support Duration (FOSD) within 14 Days of Enrollment | 14 days of enrollment
The Impact of HDIVC on Early Inflammatory Markers in SAP, Including the Levels and Changes of C-Reactive Protein and Inflammatory Cytokines IL-6, IL-1, and IL-10 | 28 days of enrollment
the Duration of Systemic Inflammatory Response Syndrome (SIRS) | 28 days of enrollment
  The scoring system primarily includes the following four clinical indicators. If ≥2 criteria are met, SIRS can be diagnosed:
  1. Temperature >38°C or <36°C
  2. Heart Rate>90 beats per minute
  3. Respiratory rate >20 breaths per minute, or arterial PaCO₂ <32 mmHg
  4. Abnormal White Blood Cell (WBC) Count >12×10⁹/L or <4×10⁹/L, or immature neutrophils >10%
The Impact of HDIVC on Sequential Organ Failure Assessment (SOFA) Score | 28 days of enrollment
  The SOFA score involves six major organ systems, including the respiratory system, hematologic system (platelets), liver function, renal function, central nervous system, and circulatory system (blood pressure). Each system is scored from 0 to 4, with a total score ranging from 0 to 24. Higher scores indicate that the organ failure is more severe.
The Impact of HDIVC on Modified Marshall Score | 28 days of enrollment
  This scoring system primarily evaluates three key organ systems (respiratory system, circulatory system and renal function), with each system scored from 0 to 4. If any system scores ≥2, organ dysfunction is considered present.
The Impact of HDIVC on Fluid Retention | 28 days of enrollment
  assessment of fluid retention, defined as the total input volume of intravenous fluid and enteral nutrition minus the output volume of urine and drainage
The Impact of HDIVC on Acute Physiology and Chronic Health Evaluation II (APACHE II) Score | 28 days of enrollment
  It is a severity-of-disease classification system used to assess critically ill patients and predict hospital mortality. The score is calculated based on three main components: Acute Physiology Score (APS) (0-60 points), Age Score (0-6 points) and Chronic Health Condition Score (0-5 points). It has a maximum total score of 71 points. The higher the APACHE II score, the greater the risk of mortality.
The Impact of HDIVC on Bedside Index for Severity in Acute Pancreatitis (BISAP) Score | 28 days of enrollment
  It is a scoring system used for early assessment of disease severity and prognosis in patients with acute pancreatitis (AP). Each item scores 1 point, total 0-5 points.
  B - BUN > 25 mg/dL (Blood Urea Nitrogen > 25 mg/dL) I - Impaired mental status (Glasgow Coma Scale [GCS] < 15) S - SIRS (Systemic Inflammatory Response Syndrome) (Meeting ≥2 criteria) A - Age > 60 years P - Pleural effusion BISAP helps predict mortality risk and complications.0-1 points means very low mortality risk (<1%). 2-3 points means moderate risk (mortality rate ~2-10%). 4-5 points means high risk (mortality rate >20%).
The Impact of HDIVC on Pancreatic Necrosis, namely Computed Tomography Severity Index (CTSI). | 28 days of enrollment
  It is a scoring system used to assess the severity of acute pancreatitis (AP) based on contrast-enhanced CT (CECT) imaging. CTSI helps predict disease severity, complications, and prognosis. It categorizes acute pancreatitis severity as follows:
  0-3 points: Mild pancreatitis, low risk of complications 4-6 points: Moderate pancreatitis, higher risk of complications and organ failure 7-10 points: Severe pancreatitis, high risk of necrosis, organ failure, and mortality
The Incidence of IPN (Infection-Related Pancreatic Necrosis) | 28 days of enrollment
ICU Stay Duration | through study completion, an average of 6 months
Hospitalization Costs | through study completion, an average of 6 months
Plasma Concentration of Vitamin C Before and After Treatment | 28 days of enrollment
Adverse events related to Vitamin C | 28 days of enrollment
The Impact of HDIVC on the Composition of the Gut Microbiota | 28 days of enrollment
  The study use the fecal sample to assess the composition of gut microbiota using sequencing techniques (16S rRNA, metagenomics), diversity analysis (alpha and beta diversity), functional profiling (metabolomics) and inflammation markers (calprotectin).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Jiao Tong University School of Medicine Affiliated Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No